CLINICAL TRIAL: NCT07126834
Title: Could a Breathing Protocol Serve as a Non-Pharmacological Strategy to Mitigate Acute Mountain Sickness? A Randomized Crossover Trial.
Brief Title: Voluntary Isocapnic Hyperpnea in Hypoxia to Mitigate Acute Mountain Sickness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Sport - National Research Institute, Poland (Other)
Responsible Party: Principal Investigator, Tomasz Kowalski, Principal Investigator - Research Associate, Institute of Sport - National Research Institute, Poland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025/TK/1; 102.39/2025 (Other Grant/Funding Number: Institute of Sport-National Research Institute, Poland)
Record Dates: First submitted 2025-08-06; First posted 2025-08-17 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Mountain Sickness
Keywords: acute mountan sickness; breathing; hyperpnoea; blood gas analysis; lake louis scale
MeSH Terms: conditions — Altitude Sickness; Respiratory Aspiration; Hyperventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Across 2 consecutive days, the participants underwent two 2-hour sessions under hypoxia of 4200m asl (FiO2 = 12.8%) in a normobaric chamber (Air Sport, Międzyzdroje, Poland). The sessions were held at the same time of day, between 17:00 and 19:00. Temperature (approximately 21 °C), humidity (45-50%), and gas concentration were centrally controlled and maintained at stable levels throughout the exposure period. During the control session, the participants remained seated without any activity.
- Experimental (Experimental): Across 2 consecutive days, the participants underwent two 2-hour sessions under hypoxia of 4200m asl (FiO2 = 12.8%) in a normobaric chamber (Air Sport, Międzyzdroje, Poland). The sessions were held at the same time of day, between 17:00 and 19:00. Temperature (approximately 21 °C), humidity (45-50%), and gas concentration were centrally controlled and maintained at stable levels throughout the exposure period. During the experimental session, they additionally performed a 5-minute VIH session (20 breaths/minute) after 1 hour of hypoxic exposure. Isocapnic BreathWayBetter devices (Isocapnic Technologies Inc., Kelowna, British Columbia, Canada) equipped with 6-liter breathing bags were employed to perform VIH. The accompanying Isocapnic mobile app was used to guide breathing rhythm and monitor session duration.
  Interventions: Behavioral: VIH

INTERVENTIONS:
Behavioral: VIH — During the experimental session, they additionally performed a 5-minute VIH session (20 breaths/minute) after 1 hour of hypoxic exposure. Isocapnic BreathWayBetter devices (Isocapnic Technologies Inc., Kelowna, British Columbia, Canada) equipped with 6-liter breathing bags were employed to perform VIH. The accompanying Isocapnic mobile app was used to guide breathing rhythm and monitor session duration.
  Arms: Experimental

SUMMARY:
This study investigates the effects of a brief Voluntary Isocapnic Hyperpnoea (VIH) on Acute Mountain Sickness (AMS) symptoms, SpO₂, blood pressure, and blood gas homeostasis in normobaric hypoxia, to evaluate whether such respiratory modulation may serve as a viable strategy to alleviate AMS symptoms. The investigation seeks to explore the physiological mechanisms underlying VIH in severe hypoxia (4200m asl) and furnish insight regarding practical means of providing immediate relief from AMS symptoms. Furthermore, given the scarcity of relevant literature, this investigation may serve as a pilot study and lay the foundation for future research.

The present investigation employed a randomized crossover design. The study was conducted in the Institute of Sport - National Research Institute in Warsaw, Poland, in July and August 2025. Across 2 consecutive days, the participants underwent two 2-hour sessions under hypoxia of 4200m asl (FiO2 = 12.8%) in a normobaric chamber (Air Sport, Międzyzdroje, Poland). The sessions were held at the same time of day, between 17:00 and 19:00. Temperature (approximately 21 °C), humidity (45-50%), and gas concentration were centrally controlled and maintained at stable levels throughout the exposure period. During the control session, the participants remained seated without any activity. During the experimental session, they additionally performed a 5-minute VIH session (20 breaths/minute) after 1 hour of hypoxic exposure. Isocapnic BreathWayBetter devices (Isocapnic Technologies Inc., Kelowna, British Columbia, Canada) equipped with 6-liter breathing bags were employed to perform VIH. The accompanying Isocapnic mobile app was used to guide breathing rhythm and monitor session duration. The order of sessions was determined using block randomization within subgroups of 4-6 individuals to ensure balanced exposure to each condition. Multiple measurements were taken, including blood pressure, heart rate, SpO2, blood gasometry, and the 2018 Lake Louise AMS Score.

DETAILED DESCRIPTION:
Blood gas analysis was conducted using a Radiometer™ ABL90 FLEX (Radiometer Medical ApS, Brønshøj, Denmark). The following parameters were assessed: hydrogen ion concentration (pH), bicarbonate ion concentration (HCO₃-), partial pressure of oxygen (pO₂), and partial pressure of carbon dioxide (pCO₂). All measurements were taken in duplicate using 45 µL capillary blood samples collected from the fingertip. Analyses were performed immediately following collection by a trained technician following the manufacturer's instructions.

Peripheral blood pressure was measured digitally using the OMRON M2 monitor (OMRON Healthcare, Kyoto, Japan).

SpO₂ was estimated at the fingertip using a pulse oximeter (NONIN Onyx Vantage 9590, Nonin Medical, Inc., Plymouth, MN, USA).

The 2018 Lake Louise AMS Score questionnaire was presented to the participants before the experiment for familiarization and then used to evaluate symptoms of AMS based on a combination of subjective self-reports and clinical findings.

All the measurements were performed by qualified and experienced specialists. The participants were blinded to the obtained results, except for the 2018 Lake Louise AMS Score, which was self-reported.

ELIGIBILITY:
The inclusion criteria comprised:

* age between 18 and 39 years,
* meeting the World Health Organization's minimum physical activity guidelines, defined as 150-300 minutes of moderate-intensity aerobic activity per week, 75-150 minutes of vigorous-intensity activity, or an equivalent combination of both (Bull et al. 2020).

Exclusion criteria included:

* exposure to hypoxia within the past three months,
* any chronic or acute medical condition within the same timeframe,
* current use of any medication,
* known allergic reactions,
* pregnancy,
* smoking.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
SpO₂ | Day 1 and Day 2 of the study.
  Arterial oxygen saturation (SpO₂)
AMS LL | Day 1 and Day 2 of the study.
  2018 Lake Louise Acute Mountain Sickness Score
pH | Day 1 and Day 2 of the study.
  hydrogen ion concentration
pO₂ | Day 1 and Day 2 of the study.
  partial pressure of oxygen (pO₂)
pCO₂ | Day 1 and Day 2 of the study.
  partial pressure of carbon dioxide (pCO₂)
HCO₃- | Day 1 and Day 2 of the study.
  bicarbonate ion concentration (HCO₃-)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sport - National Research Institute, Warsaw, Poland, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No
Privacy reasons.